CLINICAL TRIAL: NCT04429386
Title: Brain Responses Associated With Ingestive Behavior in Obese Women: the Effects of Bariatric Surgery, and Their Association With Behavioral, Satiety Signal Responses and Weight Loss
Brief Title: Brain Gut Axis Changes After Bariatric Surgery and Their Relationship to Weight Loss
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#13-001552
Record Dates: First submitted 2020-05-06; First posted 2020-06-12 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples for 16S RNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — Laparoscopic bariatric surgery including gastric bypass and sleeve gastrectomy

SUMMARY:
Assessing the changes in the brain-gut axis after weight loss surgery and their relationship with weight loss and changes in eating behaviors.

Obese women undergoing weight loss surgery will be recruited to participate in the study. These individuals will undergo a screening visit and 4 study visits. The study visits will occur before, and at 1-, 6- and 12 months after the weight loss surgery. Each study visit will include evaluation of brain function (fMRI), anthropometrics, blood and stool samples and eating behaviors questionnaires.

DETAILED DESCRIPTION:
Assessing the changes in the brain-gut axis after weight loss surgery and their relationship with weight loss and changes in eating behaviors.

Obese women undergoing weight loss surgery will be recruited to participate in the study. These subjects will undergo a screening visit and 4 study visits. The study visits will occur before, and at 1-, 6- and 12 months after the weight loss surgery. Each study visit will include evaluation of brain function (fMRI), anthropometrics, blood samples (gut hormones, cytokines, metabolomics ) and stool samples (16S RNA and Metabolomics) and eating behaviors questionnaires (YFAS, TFEQ, food cravings/preferences scales, 3-day food food intake records)

Primary outcomes: weight loss after surgery and changes in eating behaviors scales (YFAS, TFEQ) , metabolomics, appetite related hormones and gut microbiome (16S RNA) Secondary outcomes: changes in brain function (fMRI/MRS), diet (3-day food intake records) and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Women, age 18-55 years
* Eligible and approved for undergoing laparoscopic gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) following the Guidelines for Clinical application of Laparoscopic Bariatric Surgery by of American Gastrointestinal and Endoscopic Surgeons (SAGES)
* Right-handed

Exclusion Criteria:

* Previous major gastrointestinal surgery including weight loss surgery (partial or complete resection of stomach and/or small bowel, Whipple procedure, etc)
* Use of medications known to affect hunger, satiety, or intestinal motility.
* Unwillingness or inability to give informed consent
* Any contraindication to undergo MRI
* Current or past alcohol or drug abuse problem or smoking
* Pregnancy, lactating or post partum less than 12 months
* Body weight at enrollment greater than 350 lbs.
* Current use of insulin and or insulin dependent diabetes
* Renal insufficiency, retinopathy, or neuropathy.
* Post menopausal (defined as no menses for 12 consecutive months)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will include obese women undergoing bariatric surgery as part of standard medical care.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-02-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Percentage of excess weight loss at 6 months | Measured at 6-months after bariatric surgery
  Measure of weight loss, it is calculated using the following formula: preoperative weight - weight at the follow-up visit)/(preoperative weight - Ideal body weight *100. Greater values mean greater weight loss (better).
Percentage of excess weight loss at 12 months | Measured at 12-months after bariatric surgery
  Measure of weight loss, it is calculated using the following formula: preoperative weight - weight at the follow-up visit)/(preoperative weight - Ideal body weight *100. Greater values mean greater weight loss (better). Greater values are better.
Change in Yale Food Addiction Scale score at 6 months | Measured at baseline and at 6-months after the bariatric surgery
  Yale Food Addiction Scale that is a 25-item measure developed to measure food addiction. Score range: 0 to 7. Higher scores in the scale mean more symptoms resembling food addiction (worse).
Change in Yale Food Addiction Scale score at 12 months | Measured at baseline and at 12-months after the bariatric surgery
  Yale Food Addiction Scale that is a 25-item measure developed to measure food addiction. Score range: 0 to 7. Higher scores in the scale mean more symptoms resembling food addiction (worse).
Change in Three-Factor Eating Questionnaire score at 6-months | Measured at baseline and 6-months after the bariatric surgery
  Three-Factor Eating Questionnaire is a validated scale that is designed to measure 3 dimensions of human eating behavior: cognitive restraint of eating (Factor I), disinhibition (Factor II), and hunger (Factor III). The minimum score for factors I-II-III is therefore 0-0-0, and maximum possible score is 20-16-15. Higher scores in the respective scales are indicative of greater cognitive restraint (better), uncontrolled (worse), or emotional eating (worse).
Change in Three-Factor Eating Questionnaire score at 12-months | Measured at baseline and 12-months after the bariatric surgery
  Three-Factor Eating Questionnaire is a validated scale that is designed to measure 3 dimensions of human eating behavior: cognitive restraint of eating (Factor I), disinhibition (Factor II), and hunger (Factor III). The minimum score for factors I-II-III is therefore 0-0-0, and maximum possible score is 20-16-15. Higher scores in the respective scales are indicative of greater cognitive restraint (better), uncontrolled (worse), or emotional eating (worse).
Change in diet (3-day food intake record) at 6-months. | Measured at baseline and at 6-months after the bariatric surgery
  3-day food intake record: individuals will record everything they eat and drink for 3 days. To assess calorie intake and macro nutrients
Change in diet (3-day food intake record) at 12-months. | Measured at baseline and at 12-months after the bariatric surgery
  3-day food intake record: individuals will record everything they eat and drink for 3 days. To assess calorie intake and macro nutrients
Changes in blood levels of Ghrelin at 6-months | Measured at baseline and at 6-months after the bariatric surgery
  Serum levels of Ghrelin. Units of gut hormones include Ghrelin in pg/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of Ghrelin at 12-months | Measured at baseline and at 12-months after the bariatric surgery
  Serum levels of Ghrelin. Units of gut hormones include Ghrelin in pg/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of glucagon-like peptide (GLP)-1 at 6-months | Measured at baseline and at 6-months after the bariatric surgery
  Serum levels of glucagon-like peptide (GLP)-1. Units of gut hormones include GLP-1 in pmol/L. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of glucagon-like peptide (GLP)-1 at 12-months | Measured at baseline and at 12-months after the bariatric surgery
  Serum levels of glucagon-like peptide (GLP)-1. Units of gut hormones include GLP-1 in pmol/L. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of Peptide YY at 6-months | Measured at baseline and at 6-months after the bariatric surgery
  Serum levels of peptideYY(PYY). Units of Peptide YY in pg/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of Peptide YY at 12-months | Measured at baseline and at 12-months after the bariatric surgery
  Serum levels of peptideYY(PYY). Units of Peptide YY in pg/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of insulin at 6-months | Measured at baseline and at 6-months after the bariatric surgery
  Serum levels of insulin. Units of gut hormones include insulin in ulu/L. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of insulin at 12-months | Measured at baseline and at 12-months after the bariatric surgery
  Serum levels of insulin. Units of gut hormones include insulin in ulu/L. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of leptin at 6-months | Measured at baseline and at 6-months after the bariatric surgery
  Serum levels of leptin. Units of gut hormones include Leptin in ng/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in blood levels of leptin at 12-months | Measured at baseline and at 12-months after the bariatric surgery
  Serum levels of leptin. Units of gut hormones include Leptin in ng/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of these hormones.
Changes in gut microbiome at 6 months | Measured at baseline and at 6-months after the bariatric surgery
  High-Throughput Microbiome Sequencing for sequencing of the 16S ribosomal RNA. Output sequences are classified as domain, phylum, family and genus to species, depending on the depth of reliable classifier assignments ribosomal RNA (rRNA) gene as the genetic marker to study bacterial phylogeny and taxonomy.
Changes in gut microbiome at 12 months | Measured at baseline and at 12-months after the bariatric surgery
  High-Throughput Microbiome Sequencing for sequencing of the 16S ribosomal RNA. Output sequences are classified as domain, phylum, family and genus to species, depending on the depth of reliable classifier assignments ribosomal RNA (rRNA) gene as the genetic marker to study bacterial phylogeny and taxonomy.

SECONDARY OUTCOMES:
Changes in Brain function as measured by functional magnetic resonance imaging ( fMRI) at 6 months | Measured at baseline and at 6-months after the bariatric surgery
  Functional brain images will be obtained using established acquisition protocols for resting state and evoked brain responses
Changes in Brain function as measured by functional magnetic resonance imaging ( fMRI) at 12 months | Measured at baseline and at 12-months after the bariatric surgery
  Functional brain images will be obtained using established acquisition protocols for resting state and evoked brain responses
Changes in Inflammatory markers at 6 months | Measured at baseline and at 6-months after the bariatric surgery
  Serum levels of adipokines and inflammatory cytokines. Units include: Adiponectin in pg/ml, Interleukin 1β in pg/ml , Interleukin 6 in pg/ml, Lipopolysaccharide in pg/ml, tumor-necrosis-factor TNF-α in pg/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of adipokines and inflammatory cytokines
Changes in Inflammatory markers at 12 months | Measured at baseline and at 12-months after the bariatric surgery
  Serum levels of adipokines and inflammatory cytokines. Units include: Adiponectin in pg/ml, Interleukin 1β in pg/ml , Interleukin 6 in pg/ml, Lipopolysaccharide in pg/ml, tumor-necrosis-factor TNF-α in pg/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of adipokines and inflammatory cytokines
Changes in metabolite concentrations at 6 months. | Measured at baseline and at 6-months after the bariatric surgery
  Differences in blood metabolite concentrations measured by mass spectrometry, comparing metabolite concentrations from obese patients at baseline and after bariatric surgery.
Changes in metabolite concentrations at 12 months. | Measured at baseline and at 12-months after the bariatric surgery
  Differences in blood metabolite concentrations measured by mass spectrometry, comparing metabolite concentrations from obese patients at baseline and after bariatric surgery.

IPD SHARING:
Plan to Share IPD: Undecided